CLINICAL TRIAL: NCT05061888
Title: Using the FoodImageTM App to Assess Smart Interventions Designed to Improve Nutrition & Reduce Food Waste
Brief Title: Free Living Food Waste Management and Diet Quality Improvement Using Smart Intervention and Food Image Application
Acronym: FoodImage2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 2021-015
Record Dates: First submitted 2021-09-09; First posted 2021-09-30 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Diet, Healthy
Keywords: Food Waste; Diet Quality; Stress Management; Food Intake
MeSH Terms: interventions — Fruit; Vegetables; Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food Waste Intervention Group (Active Comparator): This group will receive an intervention on food waste management and fruit and vegetable replacement to increase diet quality while avoiding an increase in calories. Both groups will obtain free fruit and vegetable boxes and will use the FoodImage app to record food acquisition (Shop), food prep (Prep), intake (Eat) and waste (Toss) for approximately 3 (24 hour) days; ideally including 1 weekend date.
  Interventions: Other: Smart Intervention for Food Waste Management and Replacing current diet with Fruits and Vegetables
- Stress Management Control Group (Placebo Comparator): This group will receive an intervention on Stress Management and will be intensity matched to the treatment group. Both groups will obtain free fruit and vegetable boxes and will use FoodImage to record food acquisition (Shop), food prep (Prep), intake (Eat) and waste (Toss) for approximately 3 (24 hour) days; ideally including 1 weekend date.
  Interventions: Other: Smart Intervention for Stress Management

INTERVENTIONS:
Other: Smart Intervention for Food Waste Management and Replacing current diet with Fruits and Vegetables — Will receive a Smart Intervention on Food Waste Management and replacing less healthy foods with fruits and vegetables.
  Other Names: Treatment Group
  Arms: Food Waste Intervention Group
Other: Smart Intervention for Stress Management — Will receive a Smart Intervention on stress management practices and strategies.
  Other Names: Control Group
  Arms: Stress Management Control Group

SUMMARY:
The primary aim of this study is to reduce household food waste and improve individual nutrition. This will be achieved using the FoodImageTM smartphone app 1, a novel method for measuring household food acquisition, food intake, and food waste decisions, to assess the efficacy of a smart intervention that targets food waste reduction and diet quality improvement. The intervention is designed to improve nutrition by offsetting intake of less nutritious foods with increased fresh fruit and vegetable (FV) intake while simultaneously reducing household food waste via strategies tailored to participating households.

DETAILED DESCRIPTION:
Data collected will be used to:

1. Test the effects of free FV provision on: (a) household food waste levels, (b) total FV acquisition (free FV provision plus purchases post-intervention vs. pre-intervention FV purchases), and (c) the consumption of FV (Food Patterns Equivalents Database, FPED). We hypothesize that free FV provision will increase food waste, total FV acquisition, and diet quality (increase the Healthy Eating Index [HEI]). We will test these hypotheses by comparing baseline and follow-up data from participants randomly assigned to the control condition, which features free FV provision and a placebo (stress management) intervention not focused on food waste. Exploratory analyses will examine the effects on dietary energy intake and if the freely provided FV replace non-FV foods in the baseline diet.
2. Test if a smart intervention to reduce food waste and replace less healthy foods with FV significantly reduces post-intervention food waste compared to the control group while increasing FV acquisition and consumption compared to pre-intervention baseline. We hypothesize that this smart intervention will increase total FV acquisition and FV consumption compared to baseline, and these increases are not expected to differ significantly from control. It is further hypothesized that those receiving the smart intervention will significantly reduce food waste compared to controls. Exploratory analyses will examine the extent to which the smart intervention had the intended effect of replacing less healthy foods with FV consumption.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-62 years
* Body mass index (BMI) 18.5 - 50 kg/m2, based on self-reported height and weight
* Ownership of an iPhone, which the participant is willing to use for the study
* Access to Apple ID, password, and email address and willing to use them in the course of the study
* Performs a majority of household food shopping and preparation
* If children are present in household, all children are between 6-18 years
* Able to meet the schedule demands for the study

Exclusion Criteria:

* Not able to use an iPhone
* Refusal or unable to use the smartphone app to collect data in free-living conditions
* Households that purchase groceries less than 1 time per week
* More than 2 children living in the household
* Pennington Biomedical Research Center employee
* Unwilling to sign consent to use web screener questions for data set and analysis.

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2025-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Corby K Martin, PhD, Principal Investigator — Pennington Biomedical
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Stress Management Control Group: This group will receive an intervention on Stress Management and will be intensity matched to the treatment group. Both groups will obtain free fruit and vegetable boxes and will use FoodImage to record food acquisition (Shop), food prep (Prep), intake (Eat) and waste (Toss) for approximately 3 (24 hour) days; ideally including 1 weekend date.
  Smart Intervention for Stress Managment: Will receive a Smart Intervention on stress management practices and strategies.
Period: Overall Study
Arm/Group | Food Waste Intervention Group | Stress Management Control Group
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Food Waste Intervention Group | Stress Management Control Group | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (11.2) | 48.9 (11.1) | 49.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 15 | 15 | 30
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46
Fruit and Vegetable intake [Mean (Standard Deviation); unit: servings/day] — Measured using the FoodImage app, which is a validated dietary assessment method, administered at baseline and post-intervention. Fruit and vegetable intake will be quantified in servings per day, consistent with USDA dietary guidelines. At baseline and after the intervention, responses will be analyzed to determine the daily intake of fruits and vegetables.
  servings/day | 2.15 (1.5) | 2.12 (1.9) | 2.14 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: The Impact of Free FV Provision on Household FV Intake.
Description: We will test if levels of household FV intake change significantly over 4 weeks among participants randomized to the control condition, which includes free FV provision and a placebo (stress management) intervention not focused on food waste. FV intake will be measured with the FoodImage app. FV intake will be quantified as the total number of servings of FV eaten per day, with FV servings defined by United States Department of Agriculture (USDA) Food Patterns Equivalents Database (FPED).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: servings/day
Arm/Group | Food Waste Intervention Group | Stress Management Control Group
Number analyzed (Participants) | 23 | 23
servings/day | 0.72 (1.67) | -0.08 (1.34)

2. Primary Outcome: The Impact of Free FV Provision on Levels of Household Food Waste, Measured in Grams.
Description: We will test if levels of household food waste change significantly over 4 weeks among participants randomized to the control condition, which includes free FV provision and a placebo (stress management) intervention not focused on food waste. Food waste will be measured with the FoodImage app. Food waste will be quantified as total grams of food waste per day.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: grams/day
Arm/Group | Food Waste Intervention Group | Stress Management Control Group
Number analyzed (Participants) | 23 | 23
grams/day | 103.3 (253.8) | 191.0 (309.3)

3. Primary Outcome: The Impact of Free FV Provision on Levels of Household Food Waste, Measured in Calories.
Description: We will test if levels of household food waste change significantly over 4 weeks among participants randomized to the control condition, which includes free FV provision and a placebo (stress management) intervention not focused on food waste. Food waste will be measured with the FoodImage app. Food waste will be quantified as total calories of food waste per day.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Food Waste Intervention Group | Stress Management Control Group
Number analyzed (Participants) | 23 | 23
kcal/day | 101.5 (327.6) | 141.5 (316.9)

4. Primary Outcome: Change in Fruit and Vegetable Intake With Smart Intervention Compared to Pre-intervention Baseline
Description: Fruit and vegetable intake was assessed at baseline and post-intervention using data collected via the FoodImage app for three consecutive days prior to the first free fruit and vegetable pickup and three days following the final pickup. Intake was calculated in servings/day. Change is calculated as post-intervention value minus pre-intervention value, where positive values indicate an increase in intake and negative values indicate a decrease.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: servings/day
Arm/Group | Food Waste Intervention Group | Stress Management Control Group
Number analyzed (Participants) | 23 | 23
servings/day | 0.85 (0.27) | -0.07 (0.20)

5. Primary Outcome: Change in Diet Quality (Healthy Eating Index) With Smart Intervention Compared to Pre-intervention Baseline
Description: Diet quality will be assessed using the Healthy Eating Index-2020 (HEI-2020), a validated tool that measures adherence to the Dietary Guidelines for Americans. Scores range from 0 to 100, with higher scores indicating better diet quality. The total HEI score is calculated based on intake data collected via the FoodImage app over a 3-day period before and after the 4-week Smart intervention. The intervention includes the free provision of fruits and vegetables (FV) and aims to reduce food waste and replace less healthy foods with FV.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on the Healthy Eating Index
Arm/Group | Food Waste Intervention Group | Stress Management Control Group
Number analyzed (Participants) | 23 | 23
Units on the Healthy Eating Index | -2.77 (2.88) | -1.93 (1.98)

6. Primary Outcome: Determine if a Smart Intervention to Reduce Food Waste and Replace Less Healthy Foods With FV Significantly Increases FV Plate Waste Compared to Pre-intervention Baseline.
Description: We will test if levels of FV plate waste change significantly over 4 weeks among participants randomized to the control condition, which includes free FV provision and a placebo (stress management) intervention not focused on food waste. FV plate waste will be measured with the FoodImage app. FV plate waste will be quantified as total grams of food waste per day.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: grams/day
Arm/Group | Food Waste Intervention Group | Stress Management Control Group
Number analyzed (Participants) | 23 | 23
grams/day | -22.2 (13.2) | 11.7 (6.9)

7. Primary Outcome: Determine if a Smart Intervention to Reduce Food Waste and Replace Less Healthy Foods With FV Significantly Reduces Household Level Food Waste, Measured in Grams, Compared to a Control Intervention.
Description: We will test if a smart intervention to reduce food waste and replace less healthy foods with FV significantly reduces food waste over 4 weeks compared to a control (stress management) intervention. Both interventions include FV provision. Food waste will be measured with the FoodImage app. Food waste will be quantified as total grams of food waste per day.
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: grams/day
Arm/Group | Food Waste Intervention Group | Stress Management Control Group
Number analyzed (Participants) | 23 | 23
grams/day | 84.87 (41.18) | 167.19 (60.8)

8. Primary Outcome: Determine if a Smart Intervention to Reduce Food Waste and Replace Less Healthy Foods With FV Significantly Reduces Household Level Food Waste, Measured in Calories, Compared to a Control Intervention.
Description: We will test if a smart intervention to reduce food waste and replace less healthy foods with FV significantly reduces food waste over 4 weeks compared to a control (stress management) intervention. Both interventions include FV provision. Food waste will be measured with the FoodImage app. Food waste will be quantified as total calories of food waste.
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: kcal/day
Arm/Group | Food Waste Intervention Group | Stress Management Control Group
Number analyzed (Participants) | 23 | 23
kcal/day | 78.23 (49.65) | 117.37 (66.33)

9. Primary Outcome: The Impact of Free FV Provision on Household FV Acquisition.
Description: We will test if levels of household FV acquisition change significantly over 4 weeks among participants randomized to the control condition, which includes free FV provision and a placebo (stress management) intervention not focused on food waste. FV acquisition will be measured with the Foodlmage app. FV acquisition will be quantified as the total number of servings of FV acquired by the household, with FV servings defined by United States Department of Agriculture (USDA) Food Patterns Equivalents Database (FPED).
Time Frame: 4 weeks
Population: The intended outcome variable could not be quantified due to the poor quality of images and receipt scans from which the outcome variable would be generated.
Arm/Group | Food Waste Intervention Group | Stress Management Control Group
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Determine if a Smart Intervention to Reduce Food Waste and Replace Less Healthy Foods With FV Significantly Increases FV Acquisition Compared to Pre-intervention Baseline.
Description: We will test if a smart intervention to reduce food waste and replace less healthy foods with FV significantly increases FV acquisition over 4 weeks. The intervention includes free provision of FV. FV acquisition will be measured with the Foodlmage app. FV acquisition will be quantified as the total number of servings of FV acquired by the household, with FV servings defined by the United States Department of Agriculture (USDA) Food Patterns Equivalents Database (FPED).
Time Frame: 4 weeks
Population: as for outcome 9
Arm/Group | Food Waste Intervention Group | Stress Management Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline through the end of the 4-week intervention period.
Description: The study involved no greater than minimal risk.
Arm/Group | Food Waste Intervention Group | Stress Management Control Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

LIMITATIONS AND CAVEATS:
The planned statistical analysis for two primary outcomes, focused on fruit and vegetable acquisition, could not be completed. It was determined that the resolution of the data images was insufficient to accurately read numerical values and acquisition details. As a result, data extraction and encoding were not possible, affecting all records. The reported values for those two outcomes reflect only the number of participants from whom data was collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT05061888/Prot_SAP_004.pdf
  • Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT05061888/ICF_003.pdf